CLINICAL TRIAL: NCT03617640
Title: The Enteric Nervous System as Modulator of Mucosal Immune Cells
Brief Title: Neuro-Immune Interactions in the Gut
Acronym: NIG
Status: Completed | Type: Observational
Sponsor: University Children's Hospital Basel (Other)
Collaborators: University Children's Hospital, Zurich (Other); Insel Gruppe AG, University Hospital Bern (Other); Kinderspital St. Gallen (Unknown); Bâtiment Hospitalier CHUV (Unknown); Universität Klinikum Heidelberg (Unknown); Luzerner Kantonsspital (Other); Hôpitaux Universitaires Genève (Unknown); Ospedale Regionale di Bellinzona e Valli (Unknown)
Responsible Party: Principal Investigator, Simone Keck, Dr. Simone Keck, University Children's Hospital Basel
Other Study IDs: EKNZ 2015-049
Record Dates: First submitted 2018-07-24; First posted 2018-08-06 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Hirschsprung's Disease Associated Enterocolitis
Keywords: enteric neuropathies; Immune cells; Nervous cells; Microbiom
MeSH Terms: conditions — Intestinal Pseudo-Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * colonic tissue
  * blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hirschsprung's disease patients: Children diagnosed with Hirschsprung's disease or Hirschsprung's disease associated enterocolitis
- control patients: Children diagnosed and treated for miscellaneous bowel diseases

SUMMARY:
Hirschsprung's disease (HD) is diagnosed shortly after birth and is characterized by the presence of megacolon. HD is caused when ganglion cells of the enteric nervous system (ENS) in the wall of the large intestine do not develop before birth. This results in a lack of gastrointestinal motility and leads to stool obstruction. It is known that ablation of enteric nerves is associated with intestinal infection and inflammation. Indeed the most severe complication in HD is Hirschsprung's associated enterocolitis (HAEC), characterized by explosive diarrhea, abdominal distension, fever and impending septic shock. Bacteria overgrowth and changes in colonic mucosal immune cell populations during HAEC suggest a possible defect in mucosal immune homeostasis. Under steady state conditions, the mucosal immune system must be tightly controlled to avoid harmful reactions against commensal flora and food antigens, while allowing protective immune responses against invading pathogens. This balance between tolerance and defense is influenced by the mucosal microenvironment, which in turn determines the phenotype and stability of mucosal immune cell populations. The goal of this project is to understand if the enteric nervous system plays a role in regulating mucosal immunity and how this might contribute to the development of HAEC.

DETAILED DESCRIPTION:
Hirschsprung's disease (HD) is diagnosed shortly after birth and is characterized by the absence of enteric nerves in parts of colon [Amiel et al.]. Following surgical correction many patients develop HD-associated enterocolitis (HAEC), a condition distinguished by intestinal inflammation resulting in abdominal distension, severe diarrhea, fever and sepsis [Demehri et al.]. The underlying factors leading to HAEC remain poorly understood and likely involve a defect in epithelial barrier, including decreased mucin production and insufficient immunoglobulin translocation. The establishment of the epithelial barrier is dependent on epithelial recognition of microbial products by innate immune receptors, like toll-like receptors (TLRs) [Peterson et al.]. TLR-dependent epithelial recognition of microflora also coordinates the immune response away from harmless commensal bacteria and towards pathogenic invaders. Both innate and adaptive effector cell functions are influenced by epithelial-derived signals. Under homeostatic conditions commensal bacteria induce anti-inflammatory cytokines in epithelial cells which trigger a tolerogenic phenotype in mucosal antigen presenting cells (APC) resulting in generation of commensal-specific regulatory T cells (Tregs) [Curotto de Lafaille et al.]. During infection, recognition of pathogenic organisms by epithelial cells leads to secretion of inflammatory cytokines thereby inducing an inflammatory APC phenotype which promotes T effector cell (Th1, Th17) generation. The enteric nervous system is directly located underneath the epithelium and controls epithelial cell function. Ablation of enteric glia cells, one of the two cell types of the ENS, in mice is associated with inflammation and enterocolitis [Cornet et al.]. In a study from 2011 Flamant and co-workers demonstrate that enteric glia cells protect from a shigella flexneri invasion by preventing lesions in the epithelial barrier mediated by the glia cell derived neurothrophic factor S-nitrosoglutathione (GSNO) [Flamant et al.]. We hypothesize that the lack of an enteric nervous system in HD patients modulates the microbial recognition of epithelial cells and thereby the phenotype of underlying mucosal APCs and effector T cells; this might be associated with the manifestation of HAEC.

ELIGIBILITY:
Inclusion Criteria:

Informed consent

Exclusion Criteria:

No signed informed consent No blood from patients with weak general state of health

Ages: 0 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: patients between 0 and 18 years undergoing bowel resection
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2015-02-28 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Phenotypic analysis of immune and nervous cell populations | 5 years
  Determining cell frequencies and subtypes using fluorescence-activated cell sorting (FACS) and FlowJo software
Expression profil | 5 years
  RNA expression profile of whole colon tissue and single cell populations
Histological analysis | 5 years
  Microscopic analysis of colonic tissue using immunofluorescence and immunohistochemistry

SECONDARY OUTCOMES:
Microbial metagenomics sequencing | 5 years
  16S/18S/ITS Amplicon
Identifying genetic defect | 5 years
  Targeted Sanger sequencing of known Hirschsprung's disease associated genes

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Holland-Cunz, Prof, Principal Investigator — University Children's Hospital Basel
Locations (8):
- Kinderchirurgie Universität Heidelberg, Heidelberg, Germany
- Switzerland (7):
  - Ospedale Regionale di Bellinzona e Valli, Bellinzona
  - Inselspital Universität Bern, Bern
  - Hôpitaux Universitaires Genève, Geneva
  - Bâtiment Hospitalier CHUV, Lausanne
  - Luzerner Kantonsspital, Lucerne
  - Kinderspital St. Gallen, Sankt Gallen
  - Kinderspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amiel J, Lyonnet S. Hirschsprung disease, associated syndromes, and genetics: a review. J Med Genet. 2001 Nov;38(11):729-39. doi: 10.1136/jmg.38.11.729. PMID 11694544
- [Background] Demehri FR, Halaweish IF, Coran AG, Teitelbaum DH. Hirschsprung-associated enterocolitis: pathogenesis, treatment and prevention. Pediatr Surg Int. 2013 Sep;29(9):873-81. doi: 10.1007/s00383-013-3353-1. PMID 23913261
- [Background] Peterson LW, Artis D. Intestinal epithelial cells: regulators of barrier function and immune homeostasis. Nat Rev Immunol. 2014 Mar;14(3):141-53. doi: 10.1038/nri3608. PMID 24566914
- [Background] Curotto de Lafaille MA, Lafaille JJ. Natural and adaptive foxp3+ regulatory T cells: more of the same or a division of labor? Immunity. 2009 May;30(5):626-35. doi: 10.1016/j.immuni.2009.05.002. PMID 19464985
- [Background] Cornet A, Savidge TC, Cabarrocas J, Deng WL, Colombel JF, Lassmann H, Desreumaux P, Liblau RS. Enterocolitis induced by autoimmune targeting of enteric glial cells: a possible mechanism in Crohn's disease? Proc Natl Acad Sci U S A. 2001 Nov 6;98(23):13306-11. doi: 10.1073/pnas.231474098. Epub 2001 Oct 30. PMID 11687633
- [Background] Flamant M, Aubert P, Rolli-Derkinderen M, Bourreille A, Neunlist MR, Mahe MM, Meurette G, Marteyn B, Savidge T, Galmiche JP, Sansonetti PJ, Neunlist M. Enteric glia protect against Shigella flexneri invasion in intestinal epithelial cells: a role for S-nitrosoglutathione. Gut. 2011 Apr;60(4):473-84. doi: 10.1136/gut.2010.229237. Epub 2010 Dec 7. PMID 21139062
- [Background] Rusmini M, Griseri P, Lantieri F, Matera I, Hudspeth KL, Roberto A, Mikulak J, Avanzini S, Rossi V, Mattioli G, Jasonni V, Ravazzolo R, Pavan WJ, Pini-Prato A, Ceccherini I, Mavilio D. Induction of RET dependent and independent pro-inflammatory programs in human peripheral blood mononuclear cells from Hirschsprung patients. PLoS One. 2013;8(3):e59066. doi: 10.1371/journal.pone.0059066. Epub 2013 Mar 18. PMID 23527089